CLINICAL TRIAL: NCT02899728
Title: A Phase II Study of Olaparib Plus Cediranib in Combination With Standard Therapy for Small Cell Lung Cancer
Brief Title: Olaparib, Cediranib Maleate, and Standard Chemotherapy in Treating Patients With Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01363; NCI-2016-01363 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-732; s16-01472; 9974 (Other: Dana-Farber - Harvard Cancer Center LAO); 9974 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2016-09-13; First posted 2016-09-14 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma
MeSH Terms: interventions — Carboplatin; cediranib; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (chemotherapy, cediranib maleate, olaparib) (Experimental): Patients receive carboplatin IV over 60 minutes or cisplatin IV over 60 minutes on day 1 and etoposide IV over 60 minutes on days 1, 2, and 3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Patients in Arm I who have stable disease, partial, or a complete response are randomized to receive maintenance therapy or no maintenance therapy. Patients in Arm II are assigned to receive maintenance therapy.
  MAINTENANCE THERAPY: Patients receive cediranib maleate PO QD and olaparib PO BID on days 1-28.
  NO MAINTENANCE THERAPY: Patients are eligible to crossover to receive treatment with cediranib maleate and olaparib upon disease progression at the treating investigator's discretion.
  Interventions: Drug: Carboplatin; Drug: Cediranib; Drug: Cediranib Maleate; Drug: Cisplatin; Drug: Etoposide; Drug: Olaparib
- Arm II (chemotherapy, cediranib maleate, olaparib) (Experimental): Patients receive treatment as in Arm I and also receive cediranib maleate PO QD on days 1-21. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive cediranib maleate PO QD and olaparib PO BID on days 1-28.
  Interventions: Drug: Carboplatin; Drug: Cediranib; Drug: Cediranib Maleate; Drug: Cisplatin; Drug: Etoposide; Drug: Olaparib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cediranib — Given PO
  Other Names: AZD2171
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281

SUMMARY:
This phase II trial studies how well olaparib, cediranib maleate, and standard chemotherapy work in treating patients with small cell lung cancer. Drugs used in chemotherapy, such as carboplatin, cisplatin, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Olaparib and cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Olaparib, cediranib maleate, and standard chemotherapy may work better in treating patients with small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of cediranib maleate (cediranib) plus olaparib as maintenance therapy, in patients with small cell lung cancer (SCLC) who have stable disease or better (non-progressive disease or non-PD) after initial therapy, leads to improved median progression-free survival (PFS), PFS is measured in months from the time of randomization to maintenance therapy (after completion of initial therapy), compared to standard therapy (no maintenance treatment.

SECONDARY OBJECTIVES:

I. To evaluate the impact of cediranib plus olaparib maintenance therapy on median overall survival (OS) in patients with SCLC who have non-PD after initial therapy.

II. To determine whether the addition of cediranib to cisplatin/carboplatin plus etoposide during initial therapy adds benefit to response rate, median PFS and median OS.

III. To assess safety and tolerability of the combination of cediranib plus olaparib during maintenance therapy.

IV. To evaluate potential biomarkers of clinical benefit to olaparib/cediranib combination, including tumor proteomic and genomic markers, and circulating levels of cytokines and angiogenic factors, that that may be associated with clinical benefit.

OUTLINE:

INITIAL THERAPY PHASE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive carboplatin intravenously (IV) over 60 minutes or cisplatin IV over 60 minutes on day 1 and etoposide IV over 60 minutes on days 1, 2, and 3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive treatment as in Arm I and also receive cediranib maleate orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

Patients in Arm I who have stable disease, partial, or a complete response are randomized to receive maintenance therapy or no maintenance therapy. Patients in Arm II are assigned to receive maintenance therapy.

MAINTENANCE THERAPY: Patients receive cediranib maleate PO QD and olaparib PO twice daily (BID) on days 1-28.

NO MAINTENANCE THERAPY: Patients are eligible to crossover to receive treatment with cediranib maleate and olaparib upon disease progression at the treating investigator's discretion.

After completion of study treatment, patients are followed up every 3-4 months for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of extensive-stage small cell lung cancer with no prior systemic treatment
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* White blood cell count (WBC) >= 3 x 10^9/L (within 28 days prior to administration of therapy)
* No features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) on peripheral blood smear (within 28 days prior to administration of therapy)
* Absolute neutrophil count >= 1,500/mcL (within 28 days prior to administration of therapy)
* Platelets >= 100,000/mcL (within 28 days prior to administration of therapy)
* Hemoglobin >= 10 g/dL with no blood transfusion within 28 days of initiation of therapy (within 28 days prior to administration of therapy)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of therapy)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 x institutional ULN, unless liver metastases are present and then =< 5 x institutional ULN is acceptable (within 28 days prior to administration of therapy)
* Creatinine clearance >= 50 mL/min (within 28 days prior to administration of therapy)
* Proteinuria - urine protein:creatinine ratio (UPC) of =< 1 OR =< 2+ proteinuria on two consecutive urinalysis/dipstick tests taken no less than 1 week apart; patients with 2+ proteinuria on dipstick must also have a UPC of =< 0.5 on 2 consecutive samples (within 28 days prior to administration of therapy)
* Ability to swallow and retain oral medication
* The effects of olaparib and cediranib on the developing human fetus are unknown; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and male patients and their partners who are sexually active must agree to use two highly effective forms of contraception in combination for the duration of study participation and for 3 months after completion of olaparib and cediranib administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Postmenopausal or evidence of non-pregnant status for women of childbearing potential as confirmed by a negative urine or serum pregnancy test within 7 days prior to the start of therapy; postmenopausal status is defined as:

  * Age >= 60 years, or
  * Age < 60 with any one or more of the conditions below:

    * Amenorrheic for >= 1 year in the absence of chemotherapy and/or hormonal treatments,
    * Luteinizing hormone and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range,
    * Radiation-induced oophorectomy with last menses > 1 year ago,
    * Chemotherapy-induced menopause with > 1 year interval since last menses,
    * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* Ability to understand and the willingness to sign a written informed consent document
* Participants must have archival tumor tissue available for analysis (minimum 20 5 um slide) or be able to undergo a baseline fresh tumor tissue biopsy
* Adequately controlled blood pressure; (defined as systolic blood pressure [SBP] of =< 140 mmHg and diastolic blood pressure [DBP] of =< 90 mmHg) on maximum of three antihypertensive medications; participants must have a blood pressure (BP) of =< 140/90 taken in the clinic or hospital setting by a medical professional within 2 weeks prior to starting on study; it is strongly recommended that participants who are on 3 antihypertensive medications be followed by a cardiologist or a primary care physician for management of BP while on study
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction; patients can be on thyroid hormone replacement medication; asymptomatic patients with elevated thyroid stimulating hormone (TSH) with normal T4/T3 are allowed to enroll, and recommended to follow with routine thyroid function test

Exclusion Criteria:

* Patients who have had major surgery or trauma within 28 days prior to entering the study; patients must have recovered from any effects of any major surgery and surgical wound should have healed prior to starting treatment
* Patients who have had radiotherapy within 14 days prior to entering the study
* Patients with a non-healing wound, fracture, or ulcer
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Common Terminology Criteria for Adverse Events [CTCAE] grade 1 or baseline, with the exception of alopecia)
* Patients who are receiving any other investigational agents
* Patients with symptomatic central nervous system (CNS) metastases or leptomeningeal carcinomatosis should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; exceptions include patients with previously-treated CNS metastases or those with are asymptomatic, subcentimeter metastases, and have no requirement for steroids or anti-seizure medication for at least one week prior to study entry; screening with CNS imaging studies (CT scan or MRI) is required
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib, cediranib, carboplatin, cisplatin, or etoposide
* Patients with a history of myelodysplastic syndrome (MDS)
* Patients with a history of acute myeloid leukemia (AML), or patients with a history of any other primary malignancy within 3 years prior to initiation of treatment on this study; exceptions include: patients with a history of malignancies (other than AML) that were treated curatively and have not recurred within 3 years prior to study entry; resected basal and squamous cell carcinomas of the skin; and completely resected carcinoma in situ of any type
* Patients with clinically significant gastrointestinal abnormalities including, but not limited to:

  * Clinically significant signs and/or symptoms of bowel obstruction within 3 months prior to starting treatment
  * History of intra-abdominal abscess within 3 months prior to starting treatment
  * History of gastrointestinal (GI) perforation within 6 months prior to starting treatment
  * Evidence of abdominal fistula within 6 months prior to starting treatment; history of abdominal fistula will be considered eligible if the fistula was surgically repaired, and there has been no evidence of fistula for at least 6 months prior to starting treatment, and patient is deemed to be at low risk of recurrent fistula
* Patients with a history of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or insufficiently treated deep venous thrombosis (DVT) within the past 3 months; Note: Participants with recent DVT who have been treated with therapeutic anti-coagulants for at least 6 weeks are eligible, with the exception of participants being treated with warfarin, which is prohibited on this study; other oral anti-coagulants may be allowed after discussion with overall principal investigator (PI), but short half-life low molecular weight heparins are strongly preferred
* Patients with evidence of active bleeding diathesis
* Patients with hemoptysis in excess of 2.5 mL within 6 weeks prior to the first dose of study medication
* Patients receiving any medications or substances that are potent inhibitors or inducers of CYP3A4 are ineligible; the required washout period for strong inhibitors is 2 weeks and at least one week for moderate inhibitors; the required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 4 weeks for other agents
* Patients requiring concomitant therapy with phenytoin, phenobarbital, carbamazepine, or valproic acid
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; specifically, patients with any of the following within 6 months prior to starting treatment are excluded:

  * Acute myocardial infarction
  * Unstable angina
  * New York Heart Association functional classification of III or IV
  * Left ventricular ejection fraction (LVEF) < lower limit of normal (LLN) per institutional guidelines, or 55%
  * Prior allogeneic bone marrow transplant or double umbilical cord blood transplantation
  * Patients with active hepatitis (B or C)
  * Patients with active pneumonitis
* Pregnant women are excluded from this study because olaparib and cediranib are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib or cediranib, breastfeeding should be discontinued if the mother is treated with olaparib or cediranib; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with olaparib and cediranib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients must be willing and able to check and record daily blood pressure readings if receiving cediranib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sands, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (24):
- United States (24):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Chemotherapy, Cediranib Maleate, Olaparib): Patients receive carboplatin IV over 60 minutes or cisplatin IV over 60 minutes on day 1 and etoposide IV over 60 minutes on days 1, 2, and 3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Patients in Arm I who have stable disease, partial, or a complete response are randomized to receive maintenance therapy or no maintenance therapy. Patients in Arm II are assigned to receive maintenance therapy.
  MAINTENANCE THERAPY: Patients receive cediranib maleate PO QD and olaparib PO BID on days 1-28.
  NO MAINTENANCE THERAPY: Patients are eligible to crossover to receive treatment with cediranib maleate and olaparib upon disease progression at the treating investigator's discretion.
  Carboplatin: Given IV
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Cisplatin: Given IV
  Etoposide: Given IV
  Olaparib: Given PO
- Arm II (Chemotherapy, Cediranib Maleate, Olaparib): Patients receive treatment as in Arm I and also receive cediranib maleate PO QD on days 1-21. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive cediranib maleate PO QD and olaparib PO BID on days 1-28.
  Carboplatin: Given IV
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Cisplatin: Given IV
  Etoposide: Given IV
  Olaparib: Given PO
Period: Overall Study
Arm/Group | Arm I (Chemotherapy, Cediranib Maleate, Olaparib) | Arm II (Chemotherapy, Cediranib Maleate, Olaparib)
Started | 5 (0) | 3
Completed | 4 | 2
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemotherapy, Cediranib Maleate, Olaparib) | Arm II (Chemotherapy, Cediranib Maleate, Olaparib) | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival in Patients Who Receive Cediranib Maleate/Olaparib as Maintenance Therapy
Description: Will be compared to those receiving standard therapy. will use the intention-to-treat framework in which all patients randomized are considered recipients of their randomized assignment, regardless of treatment actually received.
Time Frame: From second randomization to documented disease progression or death from any cause, whichever occurs first, assessed up to 6 months
Population: Zero participants were analyzed because this trial was closed administratively per CTEP.
Arm/Group | Arm I (Chemotherapy, Cediranib Maleate, Olaparib) | Arm II (Chemotherapy, Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival (OS) Rate
Description: Additional sensitivity analyses will be conducted on OS to address the effect of potential crossover to olaparib/cediranib on overall survival estimates. These will include rank preserving structural failure time models.
Time Frame: From initial randomization to death from any cause, assessed up to 2 years
Population: Zero participants were analyzed because this trial was closed administratively per CTEP.
Arm/Group | Arm I (Chemotherapy, Cediranib Maleate, Olaparib) | Arm II (Chemotherapy, Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Adverse Events
Description: Assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 2 years
Population: Zero participants were analyzed because this trial was closed administratively per CTEP.
Arm/Group | Arm I (Chemotherapy, Cediranib Maleate, Olaparib) | Arm II (Chemotherapy, Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Response Rate
Description: Rates in each arm will be provided with exact 95% confidence intervals, and compared using the chi-squared test (or Fisher's exact test, as needed).
Time Frame: Up to 2 years
Population: Zero participants were analyzed because this trial was closed administratively per CTEP.
Arm/Group | Arm I (Chemotherapy, Cediranib Maleate, Olaparib) | Arm II (Chemotherapy, Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Blood-based Angiogenic and Deoxyribonucleic Acid (DNA) Repair Biomarkers
Description: Assessed by whole exome sequencing. Will be summarized using descriptive statistics.
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Frequency of Genomic Aberrations
Description: Will be assessed using McNemar's test and Fisher's exact test. More sophisticated analyses may include multivariable logistic regression modeling and/or competing risks analysis.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Circulating Free DNA
Description: Will be analyzed for association with patient demographics and/or disease characteristics using the Kruskal Wallis test.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not collected.
Arm/Group | Arm I (Chemotherapy, Cediranib Maleate, Olaparib) | Arm II (Chemotherapy, Cediranib Maleate, Olaparib)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT02899728/Prot_SAP_000.pdf